CLINICAL TRIAL: NCT07063667
Title: Artificial Intelligence Model-Assisted Accurate Diagnosis of Early-Stage Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Ratification NO: 2025（188）
Record Dates: First submitted 2025-05-25; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer, Metastatic; Artifical Intelligence
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training group
  Interventions: Other: bulid primary AI model
- verdict group
  Interventions: Other: verdict model and develop its function

INTERVENTIONS:
Other: bulid primary AI model — For the collected patient data, deep learning is used to perform feature screening on the selected or collected images, and malignant risk factors are determined by combining clinical significance. A neural network classifier is trained on the training set data. Variable selection: independent variables (breast MRI images, breast ultrasound images, indicators such as CA199, CA153, CA125, AFP/CEA, etc.), dependent variables (whether suffering from breast cancer and breast cancer subtypes), and the verification accuracy standard is set as the pathological biopsy result.
  Groups: training group
Other: verdict model and develop its function — The accuracy of a breast cancer prediction model is typically evaluated using multiple metrics that assess its performance in different aspects
  Groups: verdict group

SUMMARY:
Retrospectively collect the clinical data, breast MRI images, breast ultrasound images and reports, laboratory indicators (such as CA199, CA153, CA125, CEA/AFP), pathological diagnosis results, HE staining images, and existing immunohistochemical results (including CD8A, KPT5, GFRA1, PFKP, ER/PR percentage, Her-2 expression, Ki-67 index, etc.) of patients pathologically confirmed with or excluded from breast cancer in our center between January 2019 and December 2024. For biopsy specimens from patients diagnosed with breast cancer and immunohistochemically confirmed as HR+/Her-2+ during the same period, additional immunohistochemical staining for CD8A, KPT5, GFRA1, and PFKP should be performed, with images and results collected.

The collected basic clinical information, imaging data, pathological findings, and laboratory metrics of patients will serve as candidate inputs. Units of measurement will be standardized, and missing data will be imputed using the multiple imputation by chained equations algorithm. Data harmonization will employ the Box-Cox algorithm, while min-max scaling will be used for standardization. The adaptive synthetic sampling method with a balance ratio of 0.5 will address data imbalance. For the collected patient data, deep learning will be applied to screen features from the images, combined with clinical significance to identify malignant risk factors. A neural network classifier will be trained on the training set data, with independent variables including breast MRI/ultrasound images, CA199, CA153, CA125, AFP/CEA, etc., and dependent variables including breast cancer status and subtype. Pathological biopsy results will be set as the validation standard.

Model tuning will be conducted on the validation set to construct a breast cancer prediction model. It should be noted that as a single-center study, the results have limited generalizability. The further optimization and evaluation plan for the model involves using breast disease screening data from external centers for validation and refinement, evaluating the model's practical impact on clinical decision-making, and continuously tracking and optimizing its performance.

ELIGIBILITY:
Inclusion Criteria:

* Patients pathologically diagnosed with breast cancer or excluded from breast cancer
* Available pathological results of breast masses
* Involving diagnostic population onl

Exclusion Criteria:

* Suffering from mental disorders
* Presence of non-breast diseases during examination
* Presence of breast implants
* Undergoing non-breast surgery or having received radiotherapy/chemotherapy
* Lactating or pregnant women
* Missing data

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospectively collect the clinical data, breast MRI images, breast ultrasound images and reports, laboratory indicators (such as CA199, CA153, CA125, CEA/AEP), pathological diagnosis results, HE staining images, and existing immunohistochemical results (including CD8A, KPT5, GFRA1, PFKP, ER/PR percentage, Her-2 expression, Ki-67 index, etc.) of patients who were pathologically confirmed with breast cancer or excluded from breast cancer in our center between January 2019 and December 2024.
  For biopsy specimens from patients diagnosed with breast cancer and immunohistochemically confirmed as HR+/Her-2+ between January 2019 and December 2024, additional immunohistochemical staining for CD8A, KPT5, GFRA1, and PFKP should be performed, and the immunohistochemical images and results should be collected.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
AUC (Area Under the ROC Curve) | Baseline-AUC1 Perioperative/Periprocedural-AUC2

CONTACTS AND LOCATIONS:
Locations (1):
- Army medical Cnter, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No